CLINICAL TRIAL: NCT05952739
Title: Maternal Endocrine System and Metabolic Diseases and Offspring Health: Prediction Within a Birth Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xinhua Xiao, Chief physician, Peking Union Medical College Hospital
Other Study IDs: 2022-PUMCH-C-019
Record Dates: First submitted 2023-07-04; First posted 2023-07-19 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Thyroid Dysfunction; Diabetes Mellitus
Keywords: Hyperglycemia during pregnancy; Thyroid Dysfunction During Pregnancy; Offspring metabolic diseases
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mother's blood, milk, urine, feces, placenta, fetal umbilical cord blood, and offspring's urine, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease group: No interventions
- Control group: No interventions

SUMMARY:
The incidence of metabolic diseases in pregnant women is increasing rapidly, and the risk of metabolic diseases in children is also increasing. However, there is a lack of early predictive indicators for metabolic diseases in children, which cannot effectively prevent and treat metabolic diseases in children. This project will establish a clinical database and a long-term follow-up biological bio-bank through the follow-up of metabolic indicators before and during pregnancy, and form an early warning system for the effects of maternal endocrine and metabolic diseases on the metabolism of offspring. It will not only help to warn the impact of maternal endocrine system and metabolic diseases on the metabolism of offspring, but also build a transformation platform for the study of maternal endocrine and metabolic diseases and metabolic health of offspring, which has important clinical value for curbing the rapid growth of metabolic diseases such as diabetes and obesity in China. It is expected to provide an important theoretical basis for the window period of prevention and treatment of endocrine and metabolic diseases in China.

DETAILED DESCRIPTION:
Due to the rapid changes in the environment and lifestyle, women of childbearing age often suffer from endocrine and metabolic diseases such as diabetes and thyroid diseases, resulting in poor intrauterine development environment in the early life. Maternal endocrine metabolic diseases and nutritional status not only affect their own health, but also greatly affect the metabolic health of their offspring. Hyperglycemia and thyroid dysfunction during pregnancy can increase the risk of obesity, metabolic syndrome and diabetes in offspring. The developmental origin of health and disease (DOHaD) is a well-known theory about the effect of early developmental environment (fetus and newborn) on the metabolic health of offspring. Several well-known international birth cohorts have confirmed that maternal malnutrition during pregnancy can lead to an increased risk of metabolic diseases in adult offspring. Previously, Xiao 's team found that low birth weight was an independent risk factor for abnormal glucose and lipid metabolism in adulthood through the 'Concord birth-old age' cohort study, which confirmed the DOHaD theory for the first time in the Chinese population. The above retrospective cohort study provides epidemiological evidence for the DOHaD theory. However, due to its early start and the lack of a comprehensive database of clinical data and biological samples at different stages of the subjects' lives, it is difficult to deeply analyze the high-risk factors of metabolic abnormalities in offspring, and it is difficult to effectively intervene and block the 'origin of metabolic diseases' from the early stage of life development. In addition, cross-generational studies at home and abroad are mostly retrospective and cross-sectional studies, with selection bias and information bias. Prospective birth cohort studies covering the whole life cycle of maternal endocrine and metabolic diseases are urgently needed. This project will continue to focus on the endocrine system and metabolic diseases of women of childbearing age in this large birth cohort, and cooperate with the Department of Endocrinology, Obstetrics, Pediatrics and Nutrition of Peking Union Medical College Hospital to construct a large-scale prospective cohort of maternal endocrine and metabolic diseases in the whole pregnancy cycle, establish a clinical database and a long-term follow-up bio-bank, and form an early predictive system for the impact of maternal endocrine and metabolic diseases on the metabolism of offspring, so as to provide a scientific basis for comprehensively predicting the short-term and long-term metabolic trajectories of offspring.

ELIGIBILITY:
lnclusion Criteria:

* Pregnant women
* Voluntary signing of informed consent

Exclusion Criteria:

* Twin or multiple pregnancy
* Severe pregnancy complications
* Complicated with important heart, liver, kidney, blood system and autoimmune diseases before pregnancy
* Associated with other diseases that may affect intestinal flora or metabolomics, including inflammatory bowel disease, irritable bowel syndrome, celiac disease, etc.
* Gastrointestinal and biliary surgeries, including bariatric surgery and cholecystectomy
* History of smoking, alcoholism, narcotic drug use
* For women who keep stool samples: antibiotics within 2 months of specimen collection: probiotics within 1 week of specimen collection: take oral drugs that may affect intestinal flora.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with metabolic disease before or during pregnancy and control group
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Gestational diabetes mellitus | Measure blood glucose up to 28 weeks of pregnancy
  Hyperglycemia during pregnancy; 50 participants with hyperglycemia during pregnancy
Thyroid dysfunction during pregnancy | Measure thyroid function up to 28 weeks of pregnancy
  Slightly higher TSH or positive TPOAb; 140 participants with thyroid dysfunction during pregnancy
Abnormal metabolism of offspring | 1 year
  Abnormal birth weight，blood sugar etc; 300 participants
Diabetes mellitus complicating pregnancy | Measure blood glucose up to 28 weeks of pregnancy
  Hyperglycemia during pregnancy; 50 participants with hyperglycemia during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Xiao, Study Director — Key Laboratory of Endocrinology, Ministry of Health, Department of Endocrinology, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences, Beijing 100730, China
Locations (1):
- Key Laboratory of Endocrinology, Ministry of Health, Department of Endocrinology, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences, , China, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun H, Saeedi P, Karuranga S, Pinkepank M, Ogurtsova K, Duncan BB, Stein C, Basit A, Chan JCN, Mbanya JC, Pavkov ME, Ramachandaran A, Wild SH, James S, Herman WH, Zhang P, Bommer C, Kuo S, Boyko EJ, Magliano DJ. IDF Diabetes Atlas: Global, regional and country-level diabetes prevalence estimates for 2021 and projections for 2045. Diabetes Res Clin Pract. 2022 Jan;183:109119. doi: 10.1016/j.diabres.2021.109119. Epub 2021 Dec 6. PMID 34879977
- [Background] Osmond C, Barker DJ. Fetal, infant, and childhood growth are predictors of coronary heart disease, diabetes, and hypertension in adult men and women. Environ Health Perspect. 2000 Jun;108 Suppl 3(Suppl 3):545-53. doi: 10.1289/ehp.00108s3545. PMID 10852853
- [Background] Xiao X, Zhang ZX, Cohen HJ, Wang H, Li W, Wang T, Xu T, Liu A, Gai MY, Ying S, Schmitz O, Yi Z. Evidence of a relationship between infant birth weight and later diabetes and impaired glucose regulation in a Chinese population. Diabetes Care. 2008 Mar;31(3):483-7. doi: 10.2337/dc07-1130. Epub 2007 Dec 10. PMID 18070988
- [Background] Rawal S, Olsen SF, Grunnet LG, Ma RC, Hinkle SN, Granstrom C, Wu J, Yeung E, Mills JL, Zhu Y, Bao W, Ley SH, Hu FB, Damm P, Vaag A, Tsai MY, Zhang C. Gestational Diabetes Mellitus and Renal Function: A Prospective Study With 9- to 16-Year Follow-up After Pregnancy. Diabetes Care. 2018 Jul;41(7):1378-1384. doi: 10.2337/dc17-2629. Epub 2018 May 4. PMID 29728364
- [Background] Kooijman MN, Kruithof CJ, van Duijn CM, Duijts L, Franco OH, van IJzendoorn MH, de Jongste JC, Klaver CC, van der Lugt A, Mackenbach JP, Moll HA, Peeters RP, Raat H, Rings EH, Rivadeneira F, van der Schroeff MP, Steegers EA, Tiemeier H, Uitterlinden AG, Verhulst FC, Wolvius E, Felix JF, Jaddoe VW. The Generation R Study: design and cohort update 2017. Eur J Epidemiol. 2016 Dec;31(12):1243-1264. doi: 10.1007/s10654-016-0224-9. Epub 2017 Jan 9. PMID 28070760
- [Background] Lv H, Diao F, Du J, Chen T, Meng Q, Ling X, Li H, Song C, Xi Q, Jiang Y, Xu Y, Tao S, Huang L, Wen M, Peng M, Liu C, Lu Q, He Y, Yin Y, Liu X, Xu B, Han X, Zhou K, Jiang T, Zhao Y, Ma H, Jin G, Xia Y, Liu J, Lin Y, Hu Z, Shen H. Assisted reproductive technology and birth defects in a Chinese birth cohort study. Lancet Reg Health West Pac. 2021 Jan 22;7:100090. doi: 10.1016/j.lanwpc.2020.100090. eCollection 2021 Feb. PMID 34327418
- [Background] Wang YY, Li Q, Guo Y, Zhou H, Wang QM, Shen HP, Zhang YP, Yan DH, Li S, Chen G, Zhou S, He Y, Yang Y, Peng ZQ, Wang HJ, Ma X. Ambient temperature and the risk of preterm birth: A national birth cohort study in the mainland China. Environ Int. 2020 Sep;142:105851. doi: 10.1016/j.envint.2020.105851. Epub 2020 Jun 22. PMID 32585501
- [Background] Zhou L, Li S, Zhang Q, Yu M, Xiao X. Maternal Exercise Programs Glucose and Lipid Metabolism and Modulates Hepatic miRNAs in Adult Male Offspring. Front Nutr. 2022 Mar 1;9:853197. doi: 10.3389/fnut.2022.853197. eCollection 2022. PMID 35299765
- [Background] Liu J, Ding L, Zhai X, Wang D, Xiao C, Hui X, Sun T, Yu M, Zhang Q, Li M, Xiao X. Maternal Dietary Betaine Prevents High-Fat Diet-Induced Metabolic Disorders and Gut Microbiota Alterations in Mouse Dams and Offspring From Young to Adult. Front Microbiol. 2022 Apr 5;13:809642. doi: 10.3389/fmicb.2022.809642. eCollection 2022. PMID 35479641
- [Background] Zhang Q, Sun X, Xiao X, Zheng J, Li M, Yu M, Ping F, Wang Z, Qi C, Wang T, Wang X. The effect of maternal chromium status on lipid metabolism in female elderly mice offspring and involved molecular mechanism. Biosci Rep. 2017 Apr 28;37(2):BSR20160362. doi: 10.1042/BSR20160362. Print 2017 Apr 30. PMID 28320771
- [Background] Zhou L, Xiao X, Li M, Zhang Q, Yu M, Zheng J, Deng M. Maternal Exercise Improves High-Fat Diet-Induced Metabolic Abnormalities and Gut Microbiota Profiles in Mouse Dams and Offspring. Front Cell Infect Microbiol. 2020 Jun 17;10:292. doi: 10.3389/fcimb.2020.00292. eCollection 2020. PMID 32626663